CLINICAL TRIAL: NCT04515394
Title: A Phase II Single-Arm Study to Investigate Tepotinib Combined With Cetuximab in RAS/BRAF Wild-Type Left-Sided mCRC Patients Having Acquired Resistance to Anti-EGFR Antibody Targeting Therapy Due to MET Amplification (PERSPECTIVE)
Brief Title: Study of Tepotinib Combined With Cetuximab in Participants With Left-Sided RAS/BRAF Wild Type Metastatic Colorectal Cancer (PERSPECTIVE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to operational challenges identifying suitable participants for screening in the study.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS202202_0002; 2020-001776-15 (EudraCT Number)
Record Dates: First submitted 2020-08-11; First posted 2020-08-17 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal cancer; RAS wild-type; Tepotinib; Cetuximab; Erbitux; Epidermal growth factor receptor resistance; Hepatocyte growth factor; Panitumumab; Mesenchymal epithelial transition
MeSH Terms: conditions — Colorectal Neoplasms; Deafness, Autosomal Recessive 39 | interventions — tepotinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tepotinib + Cetuximab (Experimental)
  Interventions: Drug: Tepotinib; Biological: Cetuximab

INTERVENTIONS:
Drug: Tepotinib — Participants received Tepotinib film-coated tablets at a dose of 500 milligrams (mg) orally, once daily (QD) until disease progression (according to Response Evaluation Criteria in Solid Tumors Version 1.1 [RECIST v1.1]), death, Adverse event (AE) leading to discontinuation, study withdrawal, or withdrawal of consent, whichever occurs first.
  Other Names: MSC2156119J
Biological: Cetuximab — Participants received weekly intravenous infusions of Cetuximab at a dose of 250 milligrams per square meter (mg/m^2) until disease progression (according to Response Evaluation Criteria in Solid Tumors Version 1.1 [RECIST v1.1]), death, Adverse event (AE) leading to discontinuation, study withdrawal, or withdrawal of consent, whichever occurs first.
  Other Names: Erbitux®; MSB0010442D

SUMMARY:
The purpose of this study was to assess the preliminary antitumor activity, safety and tolerability of tepotinib in combination with cetuximab in participants with RAS/BRAF wild-type left-sided Metastatic Colorectal Cancer (mCRC) having acquired resistance to anti-epidermal growth factor receptor (EGFR) antibody targeted therapy due to mesenchymal epithelial transition (MET) amplification.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (locally advanced or metastatic) left sided (from splenic flexure to rectum - National Comprehensive Cancer Network [NCCN] version 4.2020) colorectal cancer (CRC) with RAS/BRAF wild-type at study entry confirmed prior to enrollment, with previous anti-epidermal growth factor receptor (anti-EGFR) therapy and acquired resistance on the most recent anti-EGFR monoclonal antibody therapy (panitumumab or cetuximab) by radiological documentation of disease progression according to RECIST Version 1.1
* Mesenchymal epithelial transition (MET) amplification detected by a positive liquid biopsy and/or tissue with appropriate regulatory status (collected after disease progression of the previous anti-EGFR therapy)
* Measurable disease by Investigator in accordance with RECIST Version 1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Life expectancy greater than 3 months
* Participants having at least one systemic treatment for mCRC including 1 anti-EGFR monoclonal antibody therapy as the most recent line of therapy for mCRC before study treatment and must have shown a radiologically confirmed by RECIST Version 1.1 complete response (CR) or partial response (PR), both for at least 4 months or stable disease (SD) for at least 6 months to that therapy prior to disease progression
* Less than 2 months between the last administration of the most recent EGFR containing regimen and first dosing in this study
* Adequate hematological function, hepatic and renal functions as defined in the protocol
* Signed and dated informed consent indicating that the participants had been informed of all the pertinent aspects of the trial prior to enrollment
* Contraceptive use by males or females will be consistent with local regulations on contraception methods for those participating in clinical studies
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS metastases. Also excluded are participants with carcinomatous meningitis
* Participants who have brain metastasis as the only measurable lesion
* Prior chemotherapy, biological therapy, radiation therapy, hormonal therapy for anti-cancer purposes, targeted therapy, or other investigational anticancer therapy (not including palliative radiotherapy at focal sites) within 21 days prior to the first dose of study intervention, except for the anti-EGFR containing regimen including associated chemotherapy if applicable, which may be continued until enrollment of the participant in the study
* Any unresolved toxicity Grade 2 or more according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0, from previous anticancer therapy excluding neuropathy, alopecia and rash
* Severe hypersensitivity reactions to monoclonal antibodies (Grade greater than or equal to [>=] 3 NCI-CTCAE v 5.0), any history of anaphylaxis, or uncontrolled asthma (i.e., 3 or more occurrences of partially controlled asthma)
* Discontinuation of the most recent cetuximab or panitumumab containing therapy due to an adverse event
* Prior treatment with other agents targeting the hepatocyte growth factor (HGF)/Mesenchymal epithelial transition (MET) pathway
* Impaired cardiac function: Left ventricular ejection fraction less than [<] 45 percent [%] defined by echocardiography (a screening assessment not required for participants without a history of congestive heart failure unless clinically indicated); Serious arrhythmia; Unstable angina pectoris; New York Heart Association heart failure Class III and IV; Myocardial infarction within the last 12 months prior to study entry and Symptomatic pericardial effusion; Corrected QT interval by Fridericia (QTcF) greater than (>) 480 milliseconds (ms)
* Hypertension uncontrolled by standard therapies (not stabilized to less than [< ]150/90 millimeter of mercury [mmHg])
* History of neoplasm other than mCRC
* History of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the test products
* Known infection with human immunodeficiency virus, or an active infection with hepatitis B or hepatitis C virus
* Major surgery within 28 days prior to Day 1 of study intervention
* History of Interstitial lung disease (ILD) or interstitial pneumonitis including radiation pneumonitis that required steroid treatment
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (65):
- United States (13):
  - Mayo Clinic, Phoenix, Arizona
  - Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles (UCLA), Santa Monica, California
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - North Shore-LIJ Monter Cancer Center, Lake Success, New York
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Scott & White Vasicek Cancer Treatment Center, Temple, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Aurora Cancer Care - Milwaukee West, Wauwatosa, Wisconsin
- Belgium (2):
  - Antwerp University Hospital, Antwerp
  - UZ Leuven, Leuven
- Czechia (4):
  - Universtity Hospital Brno, Brno
  - University Hospital Olomouc, Olomouc
  - Dept. of Oncology Faculty Hospital Motol, Prague
  - Hospital Na Bulovce, Prague
- France (8):
  - CHU Besançon Hôpital Jean Minjoz, Besançon
  - University Hospital of Besançon, Besançon
  - CHU Estaing, Clermont-Ferrand
  - CHU Hôpital Henri Mondor, Créteil
  - Clinique Victor Hugo, Le Mans
  - CHU de Poitiers, Poitiers
  - Curie Institute, Saint-Cloud
  - Institut Curie - René-Huguenin Hospital, Saint-Cloud
- Italy (10):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura die Tumori, Meldona
  - Fondazione IRCCS - Istituto Tumori Milano, Milan
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori, Fondazione G. Pascale Napoli, Napoli
  - UOC Oncoematologia AOU Vanvitelli, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana-Ospedale Santa Chiara, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - Foundation IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo FG
- Russia (12):
  - Arkangelsk Clinical Oncological Dyspensary, Arkhangelsk
  - Chelyabinsk Regional Clinical Center of Oncology and Nuclear Medicine, Chelyabinsk
  - Kursk Regional Clinical Oncology Dispensary, Kislino
  - FSBI "National Medical Research Center of Oncology n.a. N.N. Blokhina" of the MoH of the RF, Moscow
  - Limited Liability Company Medicine 24/7, Moscow
  - Russian Cancer research center n.a. N.N. Blokhin, Moscow
  - Omsk Regional Oncology Dispensary, Omsk
  - LLC Clinica UZI 4D, Pyatigorsk
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Tomsk National Research Medical Center, Tomsk
  - MKMC Medical City, Tyumen
  - SAHI Republican Clinical Oncology Dispensary, Ufa
- Spain (11):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - VHIO Valle de Hebron Instituto de Oncologia, Barcelona
  - H.U. Ramon y Cajal, Madrid
  - HM-CIOCC, Madrid
  - Hospital de Madrid Norte Sanchinarro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital UNiversitario La Paz, Madrid
  - H.U.Marqués de Valdecilla, Santander
  - HUVirgen del Rocio, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
- United Kingdom (5):
  - Bristol Oncology Centre, Bristol
  - Beatson WJSCC, Glasgow
  - Guy's & St Thomas' NHS Foundation Trust, London
  - The Royal Marsden Hospital, London
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202202_0002
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Targeting MET Clinical Trial Program — https://www.clinicaltrials.targeting-met.com/en

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 57 participants were screened. Out of which, 3 participants were enrolled and 2 participants received treatment in this study.
Groups:
- Tepotinib + Cetuximab: Participants received Tepotinib film-coated tablets at a dose of 500 milligrams (mg) orally, once daily (QD) in combination with weekly intravenous infusions of Cetuximab at a dose of 250 milligrams per square meter (mg/m^2) until disease progression (according to Response Evaluation Criteria in Solid Tumors Version 1.1 [RECIST v1.1]), death, Adverse event (AE) leading to discontinuation, study withdrawal, or withdrawal of consent, whichever occurs first.
Period: Overall Study
Arm/Group | Tepotinib + Cetuximab
Started | 3
Treated | 2
Completed | 2
Not Completed | 1
Not completed — Participant did not receive treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs) According to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: DLTs are defined as any of the following toxicities and judged by Investigator and/ Sponsor to be not attributable to the disease/disease-related processes under investigation: Grade 4 neutropenia for more than 7 days; Grade greater than or equal to [>=] 3 febrile neutropenia with absolute neutrophil count < 1000 per cube millimeter (per mm^3) and a single temperature of > 38.3 degree Celsius/a sustained temperature of >= 38 degree Celsius for more than 1 hour; Grade 4/Grade 3 thrombocytopenia with non-traumatic bleeding; Grade 3 uncontrolled nausea/vomiting and/diarrhea that has not improved within 72 hours despite adequate and optimal treatment; Grade 4 vomiting and/diarrhea; Grade >= 3 skin toxicity that has not resolved to Grade 2 after 14 days of adequate treatment; Any other Grade >= 3 non-hematological AE will be defined as DLT. Exceptions are alopecia/an isolated lipase and/amylase elevation of Grade >= 3 without clinical/radiological evidence of pancreatitis.
Time Frame: Day 1 to Day 21 of Cycle 1 (each cycle is of 21 days)
Population: DLT analysis set: all participants treated in the safety run-in period who received at least 75% of the tepotinib and cetuximab planned dose and completed the DLT period (3 weeks after start of treatment with study intervention), or who experienced a DLT during the DLT period regardless of the received amount of each study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Number of Participants With Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Investigators
Description: OR is defined as a best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all target lesions.
Time Frame: Time from first study treatment assessed up to 218 days
Population: Full analysis set (FAS) included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Investigator
Description: For participants with objective response, DoR is the time from when the complete response (CR) or partial response (PR) (whichever is first) criteria are first met until progression disease (PD) or death due to any cause within the period of 2 scheduled tumor assessments (84 or 168 days) after the last tumor assessment, whichever occurs first. PD is defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from the first dose of study drug until occurrence of PD, death due to any cause or last tumor assessment (assessed up to 218 days)
Population: None of the participants showed objective response.
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Investigators
Description: PFS is defined as the time (in months) from first administration of study intervention to the date of the first documentation of progression disease (PD) or death due to any cause within the period of 2 scheduled tumor assessments (84 or 168 days) after the last tumor assessment, whichever occurs first. PD is defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was to be estimated using Kaplan-Meier (KM) plots.
Time Frame: as for outcome 3
Population: FAS included all participants who were administered at least one dose of any study intervention.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
months | NA [NA to NA] — Median (and corresponding 95% CI) could not be estimated by KM estimates due to low sample size (2 participants) and low number of events of interest (1 participant).

5. Secondary Outcome: Overall Survival (OS) Assessed by Investigators
Description: OS is defined as the time (in months) from first administration of study intervention to the date of death. OS was to be estimated using Kaplan-Meier (KM) plots.
Time Frame: Time from first study treatment until death, assessed up to 218 days
Population: FAS included all participants who were administered at least one dose of any study intervention.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
months | NA [NA to NA] — Median (and corresponding 95% CI) could not be estimated by KM estimates as there was no event of interest (death).

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events that started or worsened after first dose of study intervention until 30 days after last dose. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs is defined as reasonably related to the study intervention.
Time Frame: Time from first study treatment up to 30 days after the last dose, assessed up to 226 days
Population: Safety analysis set (SAF) included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
Participants
  TEAEs | 2
  Treatment-related TEAEs | 2

7. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital sign assessment included assessments of height, weight, temperature, pulse rate, respiratory rate, and blood pressure. Clinical significance was determined by the investigator. Number of participants who had any clinically significant changes from baseline in vital signs were reported.
Time Frame: Time from first study treatment up to 30 days after the last dose, assessed up to 226 days
Population: SAF included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
Participants | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory investigation included hematology, biochemistry, coagulation, routine urinalysis and other screening tests (Follicle-stimulating hormone (FSH) and estradiol, Serum or highly sensitive urine human chorionic gonadotropin (hCG) pregnancy test, Serology (HIV antibody, hepatitis B surface antigen [HBsAg], and hepatitis C virus antibody) and all of the safety labs were performed locally. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in laboratory parameters were reported.
Time Frame: Time from first study treatment up to 30 days after the last dose, assessed up to 226 days
Population: SAF included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
Participants | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings included heart rate and measures PR, QRS, QT and QTcF intervals. 12-lead ECG recordings were obtained after the participants have rested for at least 5 minutes in semi-supine or supine position. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported.
Time Frame: Time from first study treatment up to 30 days after the last dose, assessed up to 226 days
Population: SAF included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
Participants | 0

10. Secondary Outcome: Number of Participants With At Least 1 Postive Anti-Drug Antibodies (ADAs) for Cetuximab
Description: Serum samples were analyzed by a validated electrochemiluminescence immunoassay method to detect the presence of antidrug antibodies (ADA). Number of participants with positive ADA were reported.
Time Frame: At Day 1 of cycle 1 (each cycle is of 21 days) and at End of Treatment (14 days after last dose, assessed up to 210 days)
Population: Immunogenicity analysis set included all participants who received at least one dose of study intervention and had at least one valid antidrug antibody (ADA) result.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Cetuximab
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Time from first study treatment up to 30 days after the last dose, assessed up to 226 days
Description: Safety analysis set (SAF) included all participants who were administered at least one dose of any study intervention.
Arm/Group | Tepotinib + Cetuximab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tepotinib + Cetuximab (N=2)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
oedema peripheral (General disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
Mucosal inflammation (General disorders) | 1
drug eruption (Skin and subcutaneous tissue disorders) | 1
paronychia (Infections and infestations) | 1
dry skin (Skin and subcutaneous tissue disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Device dislocation (Product Issues) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Weight increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04515394/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT04515394/SAP_001.pdf